CLINICAL TRIAL: NCT04699760
Title: Single-blinded, Randomized, Controlled Trial About the Effects of n-3 LCPUFAs on Weight and Functional Status in Patients With Colorectal Cancer.
Brief Title: The Effects of n-3 LCPUFAs in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2014-131
Record Dates: First submitted 2020-12-23; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Cancer Cachexia; Side Effects; Quality of Life
Keywords: cancer; nutrition; fish oil
MeSH Terms: conditions — Neoplasms | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Nutritional supplement without fish oil
  Interventions: Dietary Supplement: Placebo
- Fish oil (Active Comparator): Nutritional supplement with fish oil
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — 8 weeks, 2.2 G EPA/day
  Other Names: Smart Fish - cancer cachexia
  Arms: Fish oil
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effects of n-3 PUFAs on weight, physical funktion and quality of life in patients with colorectal cancer.

DETAILED DESCRIPTION:
Primary outcomes:

* Weight
* Physical function
* Hand-grip strength

Secondary outcomes:

* Quality of life
* Mid-upperarm circumference
* Incorporation of n-3 PUFAs into cell membranes

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Patients with diagnosed colorectal cancer with metastases treated with chemotherapy on Rigshospitalet, Copenhagen

Exclusion Criteria:

* < 18 years
* Patients in palliative care
* patients with haemophilia
* Patiens in treatment of anti-coagulation
* Patients with genetic hyperkolesterolemia
* Pre-dialytic patients (GFR<15ml/min/1,73m2 eller kreatinin ≥500 mmol/L)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | 8 weeks
  Difference in weight (kg) from inclusion to 8 week status

SECONDARY OUTCOMES:
quality of Life score | 8 weeks
  score - difference from inclusion to 8 week status (EORTC QLQ-C30 questionnaire)
Performance status - common daily abilities | 8 weeks
  combined scale - score - ADL

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Principal Investigator — University of Copenhagen
Locations (1):
- Departmen of Oncology, Rigshospital, Copenhagen, Denmark